CLINICAL TRIAL: NCT01239758
Title: An Open-Label Extension Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of ACE-031 (ActRIIB-IgG1) in Subjects With Duchenne Muscular Dystrophy
Brief Title: Extension Study of ACE-031 in Subjects With Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated based on preliminary safety data.
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A031-06
Record Dates: First submitted 2010-11-01; First posted 2010-11-11 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ACE-031 (Extension of cohort 1 from core study, A031-03) (Experimental)
  Interventions: Biological: ACE-031 (Extension of cohort 1 from core study, A031-03)
- ACE-031 (Extension of cohort 2 from core study, A031-03) (Experimental)
  Interventions: Biological: ACE-031 (Extension of cohort 2 from core study, A031-03)
- ACE-031 (Extension of cohort 3 from core study, A031-03) (Experimental)
  Interventions: Biological: ACE-031 (Extension of cohort 3 from core study, A031-03)

INTERVENTIONS:
Biological: ACE-031 (Extension of cohort 1 from core study, A031-03) — ACE-031 0.5 mg/kg subcutaneously once every 4 weeks for 24 weeks.
  Arms: ACE-031 (Extension of cohort 1 from core study, A031-03)
Biological: ACE-031 (Extension of cohort 2 from core study, A031-03) — Up to 1.0 mg/kg subcutaneously once every 2 weeks for 24 weeks.
  Arms: ACE-031 (Extension of cohort 2 from core study, A031-03)
Biological: ACE-031 (Extension of cohort 3 from core study, A031-03) — Up to 2.5 mg/kg subcutaneously once every 4 weeks for 24 weeks.
  Arms: ACE-031 (Extension of cohort 3 from core study, A031-03)

SUMMARY:
To evaluate the long-term safety and tolerability of ACE-031 administration in subjects with Duchenne muscular dystrophy (DMD) who participated in Study A031-03. [Note: This study was terminated based on preliminary safety data. Pending further analysis of safety data and discussion with health authorities, a new ACE-031 trial will be planned.]

ELIGIBILITY:
Inclusion Criteria:

* Completion of participation in Study A031-03 and Investigator approval
* Continuation of corticosteroid therapy at the same absolute dose and schedule as on Study A031-03

Exclusion Criteria:

* Participation in any other therapeutic clinical trial
* Plans to have surgery during the course of the study

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events. | From treatment initiation to End-of-Study Visit, approximately 24 weeks later.
Change in laboratory parameters and vital signs. | Baseline to End-of-Study Visit, approximately 24 weeks later.

SECONDARY OUTCOMES:
Percent change in total lean body mass by DXA scan. | Baseline to End-of-Study Visit, approximately 24 weeks later.
Percent change in total body and lumbar spine bone mineral density by DXA scan. | Baseline to End-of-Study Visit, approximately 24 weeks later.
Percent change in muscle strength score by hand-held myometry. | Baseline to End-of-Study Visit, approximately 24 weeks later.
Change in distance traveled in 6 minutes (standardized 6-Minute-Walk Test). | Baseline to End-of-Study Visit, approximately 24 weeks later.
Change in time to travel 10 meters (standardized 10-Meter-Walk/Run test). | Baseline to End-of-Study Visit, approximately 24 weeks later.
Change in pulmonary function tests. | Baseline to End-of-Study Visit, approximately 24 weeks later.

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Acceleron Investigative Site, Calgary, Alberta
  - Acceleron Investigative Site, Hamilton, Ontario
  - Acceleron Investigative Site, London, Ontario
  - Acceleron Investigative Site, Ottawa, Ontario